CLINICAL TRIAL: NCT02275078
Title: Pilot Study Evaluating the Feasibility and Potential Benefits of a Novel Approach of COPD Self-management That Includes a Phone Assessment/Reporting System (Tele-system)
Brief Title: Innovations in Treating COPD Exacerbations: Pilot Project on Action Plans Using New Technology.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jean Bourbeau, Director of the Respiratory Epidemiology and Clinical Research Unit, McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-053-BMD
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: COPD
Keywords: COPD; Action Plan; Telesystem; New technology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional (Other): The program consists of 3 components: 1) COPD self-management using an Action Plan; 2) Telesystem-Phone self-assessment/reporting system; and 3) Nurse case manager support.
  Interventions: Behavioral: COPD self-management using an action plan; Device: Telesystem-Phone self-assessment/reporting system; Other: Nurse case manager support

INTERVENTIONS:
Behavioral: COPD self-management using an action plan — Behavioral: Self-management education on the use of a self-administered prescription for exacerbation.
  Patients will be instructed to start treatment within 48 hours of experiencing an acute exacerbation of COPD and/or after starting their self-administered prescription.
Device: Telesystem-Phone self-assessment/reporting system — Phone Self-Assessment/Reporting System. The second component of the intervention is the use of a computer-linked interactive phone assessment/reporting system that can assess respiratory status and notify the nurse case manager as needed
  Other Names: Device:Interactive
Other: Nurse case manager support — Support:Nurse Case Manager Phone Support . The nurse case manager will call patients under two conditions. The first is to provide regularly scheduled follow-up education and support.The nurse case manager will also phone patients in response to answers they have provided to the phone system. i.e Worsening COPD status

SUMMARY:
The purpose of this project is to conduct a pilot study evaluating the feasibility and potential benefits of a phone assessment/reporting system (tele-system) in addition to a written action plan and nurse case manager support to improve patients' adherence to COPD treatment in those at risk for exacerbations.

Primary objective: explore the potential benefits with respect to patient's adherence, i.e., prompt use of the antibiotic and/or prednisone in the event of an exacerbation, increased adherence to maintenance medication; to increase patient's self-efficacy" in self-managing their disease; and to use more efficiently program resources, i.e., the case-manager.

Secondary objectives:

To assess the proportion of patients who effectively self manage exacerbations by using their COPD Action Plan

To assess self management of COPD patients with respect to the increased adherence to regular respiratory medication, (SmartInhaler electronic monitoring);

To assess increased self-efficacy in COPD patients identifying and managing exacerbations (baseline vs after 12 months);

To assess symptoms recovery, health status improvement, and prevention of ER visits and hospital admissions for COPD exacerbations.

To assess the efficiency in using program resources,

To evaluate the feasibility of this treatment approach and to provide pilot data (needed for a larger multi-centre clinical trial;

To evaluate the feasibility and need of assessment during and after exacerbation onset, health-related quality of life and physical activity;

To evaluate the safety of this approach; this is in terms of the delay in starting prednisone and an unfavourable outcome (ER visits and/or hospitalization).

DETAILED DESCRIPTION:
BACKGROUND: Chronic Obstructive Pulmonary Disease (COPD) is the 4th leading cause of death in Canada and the only chronic disease where mortality rates continue to climb. Acute exacerbations are common.Unfortunately, exacerbations are often viewed as trivial events or "simple bronchitis"despite being linked with accelerated lung function decline, poor health, hospital admissions and premature death.Conversely, prompt treatment reduces recovery time,improves health status, and decrease hospital admissions.In most patients, exacerbations are managed either in primary care walk-in clinics or emergency departments (ED), resulting in suboptimal management and high utilization costs.Furthermore, less severe exacerbations (~60%) remain unreported and untreated, although these likely have a significant negative impact on health. In Canada, quality indicators suggest that chronic disease management remains suboptimal, especially in COPD.

RATIONALE: In COPD clinics, the investigators group and others have shown that patients who learn how to self-monitor and manage acute exacerbations by following a COPD Action Plan have better health outcomes and lower rates of health care utilization (unplanned office visits, ED use, and hospital admissions). Key elements of effective self-management programs include a written Action Plan, standing orders for exacerbation medications (antibiotics/prednisone), and self-management skills training combined with access to nurse case manager support. However, these programs are time and resource intensive and hence very challenging to implement across practices, especially in those that are not specialized. Recent advances in patient-provider communication technology, such as interactive phone systems, show promise in helping inform and motivate patients with asthma, diabetes and hypertension to effectively self monitor symptoms and better self-manage their diseases.Communication technology offers new opportunities to develop chronic disease self-management programs that can be easily implemented and less likely to place additional burden on busy practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be adults with COPD at high risk for exacerbations
* Post bronchodilator spirometry FEV1 <80% pred. and FEV1/FVC <0.70
* Aged ≥ 40 yrs
* Smoking ≥ 10 pack-years
* 1 or more exacerbations requiring antibiotic or prednisone in the last year. (This is the population with the highest chance of having another exacerbation
* Combination therapy LABA-ICS (Advair) with or without an anticholinergic (Spiriva or Atrovent) and a rescue SABA (Ventolin)

Exclusion Criteria:

* Combination therapy LABA-ICS other than Advair
* Home oxygen for 18-24 hours/day
* Chronic CO2 retention
* Previous NIMV/MV
* Cognitive impairment
* Does not speak English or French fluently
* Severe co-morbidities such as bronchiectasis with recurrent infections, severe left congestive heart failure
* Survival <6 months
* Any significant medical condition other than COPD that may also result in dyspnea (e.g. unstable angina, BMI > 40).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10-15; Primary Completion 2016-06-08 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
- Patient adherence to action plan | within 3 days.
  Proportion of patients who initiate use of COPD Action Plan including starting exacerbation medications (i.e., antibiotics and/or prednisone) within 3 days.

SECONDARY OUTCOMES:
Respiratory medication adherence | 12 months
  Patient monitoring will be done using the SmartInhaler for Advair and Ventolin on a sample of subjects.
Self-efficacy to manage exacerbations: | 12 months
  Self-efficacy will be measured using a scale from 0-10 asking patients to rate their level of confidence, 0= not confident at all, 10=very confident, based on the "Understanding COPD questionnaire" [Wilson 2007; O'Neill 2012] and the principles of self-efficacy scale design, according to the construct proposed by Bandura.Level of confidence will be rated with respect to: taking medications as prescribed; items that are behavior-specific related to recognition and appropriate management of exacerbation including ability to identify signs of deterioration and need to initiate the prescribed action plan. CAT- The COPD Assessment Test (CAT) is a simple and quick questionnaire to give a reliable measure of health status in COPD which will complement existing approaches and will assess impact of COPD and exacerbation on the health of individual patients [Jones P 2009; Jones PW 2009].
Health care utilization | 12 months
  The Exacerbation Questionnaire provides detailed information about contacts with health care providers for both respiratory and non-respiratory problems including unplanned physician visits, Emergency Department, use and hospitalizations since the previous call. Program resources: Practice staff who assist with patient identification and chart review will be paid for their time on an hourly basis. Nurse case managers will keep records of all contact with patients (content, time spent); information on interaction between the nurse case manager and other providers (physicians, pharmacists, etc.) including type of call, who is making the call, duration and reason will be recorded.
Phone System | 12 months
  We will closely monitor use (according to symptom changes from the daily diary), record all feedback related to utilization (patients' responses using keypad vs. question verified when case manager call back the patient) and algorithm with corresponding status (Well, Worse, Alarm).

OTHER OUTCOMES:
Process and Implementation Evaluation | end of study at 12 months
  Qualitative research is the most appropriate method to explore experiences of health care providers, practice staff, study staff and patients.39 We will conduct group and individual interviews with the case manager, physicians, nurses and staff at each site. We will also interview a random sample of patients.
Covariates- Sociodemographic and clinical data | 12 months
  Information on age, sex, education, employment, marital status, living alone, BMI, weight/height, exacerbations, co-morbidities, and health resource utilization will be gathered from a questionnaire that patients complete at baseline. Smoking status will be queried and smokers will be classified as current, ex or never smoker as well and cumulative pack-years will be estimated.
Comorbidities: | 12 months
  The Charlson index40;41 a widely used indicator of comorbid conditions, will be calculated for each participant. A complete list of comorbidities will be extracted by study staff at baseline from the patient's medical chart, as well as from patient recall at the baseline visit. The global score ranges from 0 to 33, highest scores indicating more comorbidities, and was shown predictive of mortality in COPD.
Baseline respiratory status. Dyspnea will be evaluated using a 5-grade Medical Research Council (MRC) dyspnea scale. | 12 months
  Dyspnea will be evaluated using a 5-grade Medical Research Council (MRC) dyspnea scale.
Spirometry will be done according to stringent standards. Disease severity is categorized according to the GOLD classification. Measures will be obtained at baseline and end of treatment by the research coordinator. | 12 months
  will be done according to stringent standards. Disease severity is categorized according to the GOLD classification. Measures will be obtained at baseline and end of treatment by the research coordinator.
Anxiety and Depression. | 12 months
  The Patient Health Questionnaire-9 (PHQ-9) [Kroenke K, J Gen Intern Med 2001] will be used to assess and monitor depression, together with the Generalized Anxiety Disorder (GAD-7), a 7-item scale. The GAD-7 has also proved to have good sensitivity/specificity to screen for panic, social anxiety and post-traumatic stress disorder [Spitzer RL, Arch Intern Med 2006].

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourbeau, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Chest Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Farias R, Sedeno M, Beaucage D, Drouin I, Ouellet I, Joubert A, Abimaroun R, Patel M, Abou Rjeili M, Bourbeau J. Innovating the treatment of COPD exacerbations: a phone interactive telesystem to increase COPD Action Plan adherence. BMJ Open Respir Res. 2019 Apr 9;6(1):e000379. doi: 10.1136/bmjresp-2018-000379. eCollection 2019. PMID 31178998